CLINICAL TRIAL: NCT00531570
Title: Microvascular Ultrasonographic Imaging for the Detection of Early Stage Epithelial Ovarian Carcinoma
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: David Fishman, M.D., New York University School of Medicine
Other Study IDs: NYU 04-31 H11941
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Ovarian Neoplasms
Keywords: Women with ultrasound defined complex pelvic masses
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the United States, ovarian cancer is the fifth most common cancer to develop in women and causes more deaths than all other gynecologic malignancies combined. Because of the difficulties in detecting early stage ovarian cancer, 75% of women continue to be diagnosed with advanced stage disease (stage III or IV).

The National Ovarian Cancer Early Detection Program (NOCEDP) as part of the National Cancer Institute's Early Detection Research Network (EDRN) is committed to the development of effective means for the accurate detection of early stage ovarian cancer.

The last decade has seen rapid technological advances in diagnostic ultrasonography with the recent development of three-dimensional imaging.

Initial studies suggest that these new technologies improve upon the diagnostic accuracy of two-dimensional transvaginal imaging in the differentiation between benign and malignant pathology.

This improved diagnostic accuracy may promote improved patient care by separating complex benign masses from ovarian cancer therefore facilitating appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women must be greater than 21 years of age
2. Women must have a complex adnexal mass (as defined per ultrasound) which requires surgical intervention

Exclusion Criteria:

1. Known or suspected hypersensitivity to blood, blood products, or albumin.
2. Known history of congenital heart defect that creates a bi-directional or right-to-left shunt.
3. Known history of severe emphysema or a history of pulmonary emboli.
4. known history of severe pulmonary hypertension (systolic pulmonary artery pressures > 90 mmHg).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women must have a complex adnexal mass (as defined per ultrasound) which requires surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-02; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fishman, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Institute, New York, New York, United States